CLINICAL TRIAL: NCT05889065
Title: Effects of Scapular Proprioceptive Neuromuscular Facilitation on Pain and Range of Motion in Patients With Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/8
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive conventional physical therapy and the other group will receive scapular PNF with conventional physical therapy. Both groups will be recruited concurrently.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not be aware of which group the participant belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional PT Group (Active Comparator): Conventional group will receive routine physical therapy including
  10
  ultrasound(1.5w/cm2
  ,3 MHz continuous type, duration 10 minutes),hot packs (on affected region of shoulder for 10 minutes),shoulder ROM, stretching exercises, and joint mobilization five times per week for two weeks with 40 minutes duration of each session. Maitland mobilization will be given in supine position.
  · After giving glenohumeral joint distraction, caudal, dorsal, and ventral glides will be given at a rate of 2-3 oscillation/second for 1 to 2 minutes to patients. Grade I or II rhythmic oscillations will be applied in free range.
  Interventions: Procedure: Conventional Physical Therapy
- Scapular PNF + Conventional PT Group (Experimental): This group will receive scapular PNF techniques along with routine physical therapy (same as above). In this group 20 repetitions of diagonal scapular pattern (anterior elevation and posterior depression, posterior elevation and anterior depression) with 20 seconds rest period will be given to subjects. PNF techniques of rhythmic initiation and repeated contractions will be used in all patterns, applied for 40 minutes.
  Interventions: Procedure: Conventional Physical Therapy; Procedure: PNF techniques

INTERVENTIONS:
Procedure: Conventional Physical Therapy — group A will receive conventional physical therapy including
  10
  ultrasound(1.5w/cm2
  ,3 MHz continuous type, duration 10 minutes),hot packs (on affected region of shoulder for 10 minutes),shoulder ROM, stretching exercises, and joint mobilization five times per week for two weeks with 40 minutes duration of each session. Maitland mobilization will be given in supine position.
  · After giving glenohumeral joint distraction, caudal, dorsal, and ventral glides will be given at a rate of 2-3 oscillation/second for 1 to 2 minutes to patients. Grade I or II rhythmic oscillations will be applied in free range.
Procedure: PNF techniques — In this group 20 repetitions of diagonal scapular pattern (anterior elevation and posterior depression, posterior elevation and anterior depression) with 20 seconds rest period will be given to subjects. PNF techniques of rhythmic initiation and repeated contractions will be used in all patterns, applied for 40 minutes.
  Arms: Scapular PNF + Conventional PT Group

SUMMARY:
The term ''frozen shoulder'' is defined as a clinical condition with restricted active and passive range of motion (ROM) in all directions, including flexion, abduction, and rotation.The objective of the study is to determine the effects of Scapular proprioceptive neuromuscular facilitation and conventional physical therapy among patients with adhesive capsulitis.The study will be a randomized controlled trial (single-blinded parallel study), consisting of 2 groups- interventional group A and interventional group B.Group A will be given conventional physical therapy and group B will be given conventional physical therapy alongwith scapular PNF.Scapular PNF exercises are not included in our routine PT treatment programs and there is limited literature related to the PNF techniques. These techniques help develop muscular strength and endurance, joint stability, mobility, neuromuscular control and coordination all of which are aimed at improving the overall functional ability of patients.

ELIGIBILITY:
Inclusion Criteria:

* Cases diagnosed with adhesive capsulitis, both primary and secondary origin.
* Stage two and stage three of adhesive capsulitis.
* Unilateral adhesive capsulitis.
* Both males and females of the age group 40 years and above.

Exclusion Criteria:

* History of shoulder surgery or manipulation under anesthesia,
* Local corticosteroid injection administration to the affected shoulder within the last 3 months.
* Severe musculoskeletal, neurological and cardiovascular conditions.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain | 2 weeks
  Shoulder Pain will be measured on the basis of visual analogue scale of 0-100mm. A higher score signifies greater pain.

SECONDARY OUTCOMES:
Shoulder range of motion (ROM) | 2 weeks
  Shoulder range of motion (ROM) will be measured through goniometer. A higher score signifies greater range.
Scapular mobility | 2 weeks
  scapular mobility will be measured through lateral slide test (LSST)

CONTACTS AND LOCATIONS:
Overall Officials: Maryum Fatima, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan